CLINICAL TRIAL: NCT00817700
Title: Alteration of Sleep and Circadian Timing in Aging- Impact of a Sleep Debt in Middle-Aged and Older Adults
Brief Title: Impact of a Sleep Debt in Middle-Aged and Older Adults
Acronym: PPG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: #13159A; 5P01AG011412 (NIH)
Record Dates: First submitted 2009-01-05; First posted 2009-01-06 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Sleep Restriction
Keywords: Sleep; young adults; middle-age adults; older adults

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal (8 hours) sleep time (No Intervention): Subjects are studied under normal sleep time conditions.
- Sleep restriction (Experimental): Sleep restriction to 4 hours of sleep per night.
  Overnight sleep recording, measures of endocrine and metabolic (from blood), cardiovascular (measures of blood pressure and heart rate), performance ( before and after sleep restriction and after sleep recovery.
  Interventions: Other: Sleep restriction

INTERVENTIONS:
Other: Sleep restriction — Sleep restriction.
  Arms: Sleep restriction

SUMMARY:
This project has 6 aims.

1. To examine the impact of recurrent partial sleep loss in young, middle-aged and older men and women. Sleep will be restricted to 4 hours.
2. To test the hypothesis that extending bedtimes to allow for sleep recovery will reverse the metabolic, endocrine, and cardiovascular and neuro-behavioral alterations resulting from sleep restriction. Sleep will be extended to 12 hours following the 4 hour sleep restriction.
3. To test the hypothesis that there are age and gender differences in the total amount of sleep recovery obtained during the week of 12-hour bedtimes.
4. To test the hypothesis that there are age and gender differences in sleep capacity (the amount of time an individual can sleep per night when there is no sleep debt).
5. To test the hypothesis that sleep capacity is partly determined by baseline levels of slow-wave sleep and slow-wave activity.
6. To determine whether sleep capacity is related to sleep need by examining metabolic, endocrine, cardiovascular and neuro-behavioral changes with the amount of the individual sleep debt.

ELIGIBILITY:
Inclusion Criteria:

* normal weight
* healthy
* age 18-75 old

Exclusion Criteria:

* sleep disorder
* irregular life habits (shift workers, travelers)
* smokers
* on medication
* consumption of > 2 alcohol or caffeinated beverages/day

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2005-04; Primary Completion 2007-11 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Endocrine, metabolic, cardiovascular changes performance and autonomic nervous system activity before and after sleep restriction and after sleep recovery. | Completion of 23 day study

CONTACTS AND LOCATIONS:
Overall Officials: Eve Van Cauter, PhD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States